CLINICAL TRIAL: NCT00461266
Title: A Randomized, Open Label Study to Determine the Immunological Benefits of Adding Fuzeon to an Antiretroviral Regimen in HIV-infected Fuzeon-naïve Patients With Sustained HIV Viral Suppression
Brief Title: ESP Study: A Study to Assess the Effect of Adding Fuzeon (Enfuvirtide) to an Antiretroviral Regimen in Fuzeon-Naive Patients With Sustained HIV Viral Suppression.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19355
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; Antiretroviral Therapy, Highly Active

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: enfuvirtide [Fuzeon]; Drug: Antiretroviral therapy
- 2 (Active Comparator)
  Interventions: Drug: Antiretroviral therapy

INTERVENTIONS:
Drug: enfuvirtide [Fuzeon] — 90mg sc bid
  Arms: 1
Drug: Antiretroviral therapy — As prescribed

SUMMARY:
This 2 arm study will assess the immunological benefits of adding Fuzeon to an antiretroviral regimen in HIV-infected, Fuzeon-naive patients with a CD4 cell count <250 cells/mm3 and an HIV RNA viral load <400 copies/mL. Eligible patients will be randomized to receive Fuzeon 90mg bid sc in addition to their current antiretroviral therapy, or to continue their current antiretroviral therapy alone. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* documented chronic HIV infection;
* currently receiving a stable antiretroviral regimen;
* CD4 cell count <250 cells/mm3;
* HIV RNA viral load <400 copies/mL for >12 months.

Exclusion Criteria:

* prior exposure to Fuzeon;
* prior non-adherence to antiretroviral treatment regimens;
* active opportunistic infection;
* currently taking, or anticipated to take during the study, any immunomodulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean change in CD4 cell count from baseline | Week 24

SECONDARY OUTCOMES:
Change in HIV RNA from baseline | Week 24
Change in HIV RNA and CD4 cell count | Weeks 24-48
Correlation between CD4 count and HIV RNA; OIs; QoL; ADEs; SAEs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Australia (7):
  - Carlton
  - Darlinghurst
  - Melbourne
  - Miami
  - Perth
  - South Yarra
  - Sydney